CLINICAL TRIAL: NCT04518072
Title: Development of Synthetic Metabolic and Genetic Networks for the Detection of Urogenital Cancers
Brief Title: Synthetic Metabolic and Genetic Networks for Medical Diagnosics
Acronym: SynBioDiag
Status: Terminated | Type: Observational
Why Stopped: delay in erolement, decision of the sponsor
Sponsor: University Hospital, Montpellier (Other)
Collaborators: MICALIS (Unknown); CBS (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0404; 2019-A00234-53 (Other: ANSM)
Record Dates: First submitted 2020-07-01; First posted 2020-08-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Prostate; Cancer
Keywords: marker detection; blood sample
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample (1 EDTA tube, 1 Streck tube, 1 SST tube) and urine sample (100 ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biopsy prostatic group: positive biopsy (100) negative biopsy (100)
  Interventions: Other: Blood sample (1 EDTA tube, 1 SST tube, 1 Streck tube) and urine sample (100 ml)
- Control group: No prostate cancer (50)
  Interventions: Other: Blood sample (1 EDTA tube, 1 SST tube, 1 Streck tube) and urine sample (100 ml)

INTERVENTIONS:
Other: Blood sample (1 EDTA tube, 1 SST tube, 1 Streck tube) and urine sample (100 ml) — assessed biomarker in clinical samples

SUMMARY:
This is a category 3 human study, prospective, comparative, in parallel groups. A comparative qualitative and quantitative analysis of several markers in 250 samples is proposed.

DETAILED DESCRIPTION:
The assumption is that researchers can engineer synthetic metabolic and genetic networks to expand the panel of molecules that are currently known to be detected by natural systems. The investigators also hypothesize synthetic metabolic and genetic networks can be tuned for decisions making and in particular to diagnose diseases from biomarkers detections.

This project proposes for the first time a hybrid analogue / digital solution for the multiplexed detection of biomarkers using bacterial and paper-based biosensors. Biosensors can be designed using analog or digital devices. Digital devices in synthetic and natural systems are noise-resistant and useful for decision-making. Analog devices are useful for signal transmission and processing. Here the investigators take advantage of signal transmission and processing via analog transducers and adders, and then decision-making via genetic switches. Such a hybrid analogue / digital approach has not yet been developed for biosensing. Another novelty of the project is to use synthetic metabolic pathways to develop analog devices. The advantage in term of treatment, for example, consists in the fact that the speed of enzymatic reactions in an analog adder far exceeds the speed of gene expression required to create a genetic logic matrix; it becomes even more pronounced when the devices are connected in series. The methodology will be illustrated for the detection of biomarkers of prostate tumors, but it is broad enough to be applicable to other diagnoses. The choice to develop biosensors for prostate disease is of practical relevance since the current screening strategy (based on PSA measurement) can lead to overdiagnosis and cannot differentiate between patients with aggressive tumors and those with an indolent illness.This study propose to mainly develop a bacterial and paper-based biosensor system

ELIGIBILITY:
Inclusion Criteria:

* Men aged over 18
* Informed, written consent of the patient for the biological collection
* Subject affiliated to a French social security scheme or beneficiary of such a scheme

Patients specific inclusion criteria :

- Admitted to care prostate disease or suspicion of prostate cancer and with a positive or negative PSA blood result

Controls specific inclusion criteria :

- Man free from all prostate or bladder pathologies

Exclusion Criteria:

* Patient under legal protection
* Persons deprived of their liberty, protected adults or vulnerable persons
* Participants may withdraw their consent at any time and for any reason whatsoever without incurring any negative consequences without change in their usual care

Controls specific non-inclusion criteria :

* Patient with current prostatic or urinary infection
* History of treatment for prostate cancer other than surveillance management

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will compare two groups of patients with prostate cancer and controls.
Study Population: All patients admitted for prostate disease with a negative or positive PSA blood test may be included in the study if they meet the inclusion criteria.
  During the consultation, the investigator will check the eligibility of the subject against the criteria of eligibility.
  The investigator will present and explain the nature of the study so that the subject knows his rights and responsibilities, as well as the risks and possible benefits of the study. The duration of this visit will be approximately 1 hour.
  The PSA value will be collected for the group Patients-biopsy at 1 year follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Ability to detect and quantify biomarkers such as PSA in samples using biosensors platform | Up to 69 months
  The positive signal is bases on a permeation in E. coli cell membrane and recombinase switches.

SECONDARY OUTCOMES:
Investigational biomarker panel for diagnosis / Prostatic specific antigen | Baseline
  Biospecimen retention: blood serum and urine (unit mg/l)
Investigational biomarker panel for diagnosis / Creatinine | Baseline
  Biospecimen retention: blood serum and urine (unit µmol/l)
Investigational biomarker panel for diagnosis / Sarcosine | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Spermine | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Ornithine | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Choline | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis /Taurine | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Fumarate | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Serotonin | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / Putrescine | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis /ribitol | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / inositol | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis / 2-oxoglutarate | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)
Investigational biomarker panel for diagnosis /citrate | Baseline
  Biospecimen retention: blood serum and urine (unit: mg/l)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital, Montpellier, Hérault
  - Clinique Beau Soleil, Montpellier